CLINICAL TRIAL: NCT02542332
Title: Are Doctors Familiar With the Test Characteristics of Lung Cancer Screening?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Wagner Hospital (Other)
Responsible Party: Principal Investigator, Georg-Christian Funk, Priv. Doz. Dr., Otto Wagner Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Lung Cancer screening
Record Dates: First submitted 2015-08-16; First posted 2015-09-07 (Estimated); Last update posted 2015-09-07 (Estimated); Status verified 2015-08

CONDITIONS: Information About the Knowledge on the Statistical Background of Lung Cancer Screening of Doctors
Keywords: lung cancer screening; statistical background

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With Data (Active Comparator): Participants received statistical data about lung cancer screening
  Interventions: Other: With Data
- Without Data (No Intervention): Participants had no statistical data on lung cancer screening

INTERVENTIONS:
Other: With Data — The participants received statistical data about lung cancer screening in order to help them answer the questionaire
  Arms: With Data

SUMMARY:
This study evaluates whether doctors are familiar with the statistical background of lung cancer screening.

DETAILED DESCRIPTION:
Background: Screening with low-dose CT scan can prevent three deaths due to lung cancer among 1000 high-risk individuals. However, false-positive results and radiation exposure are relevant disadvantages deserving accurate consideration. Candidates for screening can only make an autonomous decision if doctors inform them correctly about the pros and cons of the method. Therefore, this study aims to evaluate, whether doctors understand the test characteristics of lung cancer screening.

Methods: In a randomized trial, 556 doctors (members of the Austrian Respiratory Society) will be invited to answer questions regarding lung cancer screening based on online case vignettes. Half of the participants will be randomized to the group 'with data' and will receive the correct solutions in advance. The group 'without data' will have to rely on prior knowledge or estimate. Primary endpoint will be the between-groups difference in the estimated number of deaths preventable by screening. Secondary endpoints will be the between-groups differences in prevalence of lung cancer, prevalence of suspicious results, sensitivity, specificity, positive-predictive value, and false negative rate. Estimations will also be compared to actual values from the literature.

ELIGIBILITY:
Inclusion Criteria:

* Doctors, who were in training or had a completed specialization training in:
* Pneumonology
* Internal Medicine
* Surgery
* or Radiology

Exclusion Criteria:

* Doctors, with a specialized training in
* ENT
* Pediatrics
* Pathology and doctors who had no e-mail address were excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2015-05; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Between-groups difference in the estimated reduction of mortality due to lung cancer screening | 14 days
  Participants had 14 days to complete the survey

SECONDARY OUTCOMES:
Between-groups difference prevalence of lung cancer | 14 days
  Participants had 14 days to complete the survey
Between-groups difference in sensitivity of lung cancer screening | 14 days
  Participants had 14 days to complete the survey
Between-groups difference in the frequency of a positive test result | 14 days
  Participants had 14 days to complete the survey
Between-groups difference in specificity of lung cancer screening | 14 days
  Participants had 14 days to complete the survey
Between-groups difference in positive predictive value of lung cancer screening | 14 days
  Participants had 14 days to complete the survey
Between-groups difference in the false negative rate of lung cancer screening | 14 days
  Participants had 14 days to complete the survey

CONTACTS AND LOCATIONS:
Overall Officials: Georg-Christian Funk, Assoc.Prof., Principal Investigator — Otto Wagner Hospital

REFERENCES:
- [Background] Couraud S, Cortot AB, Greillier L, Gounant V, Mennecier B, Girard N, Besse B, Brouchet L, Castelnau O, Frappe P, Ferretti GR, Guittet L, Khalil A, Lefebure P, Laurent F, Liebart S, Molinier O, Quoix E, Revel MP, Stach B, Souquet PJ, Thomas P, Tredaniel J, Lemarie E, Zalcman G, Barlesi F, Milleron B; French lung cancer screening statement taskforce; groupe d'Oncologie de langue francaise. From randomized trials to the clinic: is it time to implement individual lung-cancer screening in clinical practice? A multidisciplinary statement from French experts on behalf of the French intergroup (IFCT) and the groupe d'Oncologie de langue francaise (GOLF). Ann Oncol. 2013 Mar;24(3):586-97. doi: 10.1093/annonc/mds476. Epub 2012 Nov 7. PMID 23136229
- [Background] Dupont WD, Plummer WD Jr. Power and sample size calculations. A review and computer program. Control Clin Trials. 1990 Apr;11(2):116-28. doi: 10.1016/0197-2456(90)90005-m. PMID 2161310
- [Background] Gigerenzer G, Mata J, Frank R. Public knowledge of benefits of breast and prostate cancer screening in Europe. J Natl Cancer Inst. 2009 Sep 2;101(17):1216-20. doi: 10.1093/jnci/djp237. Epub 2009 Aug 11. PMID 19671770
- [Background] Herth FJ, Hoffmann H, Heussel CP, Biederer J, Groschel A. [Lung cancer screening--update 2014]. Pneumologie. 2014 Dec;68(12):781-3. doi: 10.1055/s-0034-1390899. Epub 2014 Dec 9. No abstract available. German. PMID 25489865
- [Background] Hoffrage U, Gigerenzer G. Using natural frequencies to improve diagnostic inferences. Acad Med. 1998 May;73(5):538-40. doi: 10.1097/00001888-199805000-00024. PMID 9609869
- [Background] Horeweg N, Scholten ET, de Jong PA, van der Aalst CM, Weenink C, Lammers JW, Nackaerts K, Vliegenthart R, ten Haaf K, Yousaf-Khan UA, Heuvelmans MA, Thunnissen E, Oudkerk M, Mali W, de Koning HJ. Detection of lung cancer through low-dose CT screening (NELSON): a prespecified analysis of screening test performance and interval cancers. Lancet Oncol. 2014 Nov;15(12):1342-50. doi: 10.1016/S1470-2045(14)70387-0. Epub 2014 Oct 1. PMID 25282284
- [Background] Jacobson FL, Austin JH, Field JK, Jett JR, Keshavjee S, MacMahon H, Mulshine JL, Munden RF, Salgia R, Strauss GM, Sugarbaker DJ, Swanson SJ, Travis WD, Jaklitsch MT. Development of The American Association for Thoracic Surgery guidelines for low-dose computed tomography scans to screen for lung cancer in North America: recommendations of The American Association for Thoracic Surgery Task Force for Lung Cancer Screening and Surveillance. J Thorac Cardiovasc Surg. 2012 Jul;144(1):25-32. doi: 10.1016/j.jtcvs.2012.05.059. PMID 22710038
- [Background] Jaklitsch MT, Jacobson FL, Austin JH, Field JK, Jett JR, Keshavjee S, MacMahon H, Mulshine JL, Munden RF, Salgia R, Strauss GM, Swanson SJ, Travis WD, Sugarbaker DJ. The American Association for Thoracic Surgery guidelines for lung cancer screening using low-dose computed tomography scans for lung cancer survivors and other high-risk groups. J Thorac Cardiovasc Surg. 2012 Jul;144(1):33-8. doi: 10.1016/j.jtcvs.2012.05.060. PMID 22710039
- [Background] Nuovo J, Melnikow J, Chang D. Reporting number needed to treat and absolute risk reduction in randomized controlled trials. JAMA. 2002 Jun 5;287(21):2813-4. doi: 10.1001/jama.287.21.2813. PMID 12038920
- [Background] Rasmussen JF, Siersma V, Pedersen JH, Brodersen J. Psychosocial consequences in the Danish randomised controlled lung cancer screening trial (DLCST). Lung Cancer. 2015 Jan;87(1):65-72. doi: 10.1016/j.lungcan.2014.11.003. Epub 2014 Nov 20. PMID 25433982
- [Background] Schulz C. [Lung cancer screening and management of small pulmonary nodules]. Dtsch Med Wochenschr. 2015 Mar;140(5):317-22. doi: 10.1055/s-0041-100760. Epub 2015 Mar 3. German. PMID 25734672
- [Background] Simmons J, Gould MK, Woloshin S, Schwartz LM, Wiener RS. Attitudes about low-dose computed tomography screening for lung cancer: a survey of American Thoracic Society Clinicians. Am J Respir Crit Care Med. 2015 Feb 15;191(4):483-6. doi: 10.1164/rccm.201409-1747LE. No abstract available. PMID 25679109
- [Background] Wegwarth O, Gigerenzer G. "There is nothing to worry about": gynecologists' counseling on mammography. Patient Educ Couns. 2011 Aug;84(2):251-6. doi: 10.1016/j.pec.2010.07.025. Epub 2010 Aug 16. PMID 20719463
- [Background] Wegwarth O, Schwartz LM, Woloshin S, Gaissmaier W, Gigerenzer G. Do physicians understand cancer screening statistics? A national survey of primary care physicians in the United States. Ann Intern Med. 2012 Mar 6;156(5):340-9. doi: 10.7326/0003-4819-156-5-201203060-00005. PMID 22393129
- [Result] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641
- [Derived] Schmidt R, Breyer M, Breyer-Kohansal R, Urban M, Funk GC. Do doctors understand the test characteristics of lung cancer screening? Wien Klin Wochenschr. 2018 Apr;130(7-8):238-246. doi: 10.1007/s00508-017-1305-9. Epub 2018 Jan 25. PMID 29372409